CLINICAL TRIAL: NCT02344784
Title: The Characteristics of Prepulse Inhibition in Children and Adolescents Suffering From Attention Deficit Disorder: With and Without Medication.
Brief Title: The Characteristics of Prepulse Inhibition in Children and Adolescents Suffering From Attention Deficit Disorder
Acronym: PPI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, ESSAM DAOD, Dr., HaEmek Medical Center, Israel
Other Study IDs: HaEmekMC; 0071-14 (Other: HaEmekMC)
Record Dates: First submitted 2015-01-16; First posted 2015-01-26 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Attention Deficit Disorder
Keywords: ADD; ADHD; PPI
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SR-HLAB EMG — Prepulse inhibition test using SR-HLAB EMG device will record the acoustic startle response for each participant: with and without Methylphenidate treatment
Drug: Methylphenidate — The regular daily dose of P.O methylphenidate of each participant will be given directly after the first prepulse inhibition test
  Other Names: Ritalin

SUMMARY:
The purpose of this study is to show that Prepulse inhibition test of acoustic startle response is an indicator of objective diagnostic characteristics of attention deficit disorder in children and adolescents.

by demonstrating that Prepulse inhibition test of acoustic startle response is impaired in children and adolescents suffering from attention deficit disorder in the relation to the normal function described in the literature.

The investigators will try to prove our hypothesis by an experiment that consists of two phases:

Phase I (about 25 minutes):

The patient will enter the room, will be asked to sit on a chair, and will be asked to look at a computer screen showing silent video of aquarium fish, then the patient will be connected to both the Prepulse inhibition test device and the Galvanic skin response device and pass the tests.

Phase II (about 25 minutes):

After completion of Phase I, each participant will receive his daily regular dose of methylphenidate and after an hour and a half from taking the drug, will repeat the tests, both the Prepulse inhibition test and the Galvanic skin response test.

Duration of the entire experiment is 140 minutes (two hours and twenty minutes).

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 7-18
2. Diagnosed with attention deficit hyperactivity disorder according to Diagnostic and statistical manual of mental disorders, fifth edition- Clinical diagnostic interview was performed.
3. Receive drug therapy with methylphenidate doses ranging from 0.3 mg / kg to 1 mg / kg.
4. The participant is treated with methylphenidate at least two months prior to the experiment.

Exclusion Criteria:

1. Autism.
2. Chronic neurological diseases.
3. Developmental delay.
4. Psychotic or major effective disorder (psychotic state now or in the past, schizophrenia, schizoaffective, depression, bipolar disorder)
5. Substance abuse.
6. Mental retardation.
7. Contraindicated for the treatment of methylphenidate.
8. Hearing problems.
9. Pregnancy week 20 and thereafter

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents (age 7 to 17.11 years) who are diagnosed with attention deficit hyperactivity disorder and are under the Medical surveillance of the mental health clinic for children and adolescents at the HaEmek Medical Center- Afula.
  Patients who meet the criteria for inclusion and exclusion will be offered to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-01; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Electromyography (EMG) of the right and the left Orbicularis oculi muscle will be recorded during the Prepulse inhibition test | The outcome measure will be assessed imediatly during each test and the participants will be followed for the whole duration of the experiment, an expected average of 3 hours

SECONDARY OUTCOMES:
Galvanic skin response will be measured by conductivity (Mv) units during the Prepulse inhibition test | The outcome measure will be assessed imediatly during each test and the participants will be followed for the whole duration of the experiment, an expected average of 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: AVRAHAM AVITAL, Study Chair — Technion, Israel Institute of Technology
Locations (1):
- The mental health clinic for children and adolescents at the HaEmek Medical Center, Afula, Israel

REFERENCES:
- [Background] Pastor PN, Reuben CA. Diagnosed attention deficit hyperactivity disorder and learning disability: United States, 2004-2006. Vital Health Stat 10. 2008 Jul;(237):1-14. PMID 18998276
- [Background] Faraone SV, Biederman J, Mick E. The age-dependent decline of attention deficit hyperactivity disorder: a meta-analysis of follow-up studies. Psychol Med. 2006 Feb;36(2):159-65. doi: 10.1017/S003329170500471X. PMID 16420712
- [Background] Larson K, Russ SA, Kahn RS, Halfon N. Patterns of comorbidity, functioning, and service use for US children with ADHD, 2007. Pediatrics. 2011 Mar;127(3):462-70. doi: 10.1542/peds.2010-0165. Epub 2011 Feb 7. PMID 21300675
- [Background] Biederman J, Quinn D, Weiss M, Markabi S, Weidenman M, Edson K, Karlsson G, Pohlmann H, Wigal S. Efficacy and safety of Ritalin LA, a new, once daily, extended-release dosage form of methylphenidate, in children with attention deficit hyperactivity disorder. Paediatr Drugs. 2003;5(12):833-41. doi: 10.2165/00148581-200305120-00006. PMID 14658924
- [Background] Ornitz EM, Hanna GL, de Traversay J. Prestimulation-induced startle modulation in attention-deficit hyperactivity disorder and nocturnal enuresis. Psychophysiology. 1992 Jul;29(4):437-51. doi: 10.1111/j.1469-8986.1992.tb01717.x. PMID 1410175
- [Background] Castellanos FX, Fine EJ, Kaysen D, Marsh WL, Rapoport JL, Hallett M. Sensorimotor gating in boys with Tourette's syndrome and ADHD: preliminary results. Biol Psychiatry. 1996 Jan 1;39(1):33-41. doi: 10.1016/0006-3223(95)00101-8. PMID 8719124
- [Background] Ornitz EM, Russell AT, Hanna GL, Gabikian P, Gehricke JG, Song D, Guthrie D. Prepulse inhibition of startle and the neurobiology of primary nocturnal enuresis. Biol Psychiatry. 1999 Jun 1;45(11):1455-66. doi: 10.1016/s0006-3223(98)00205-4. PMID 10356628
- [Background] Braff DL, Geyer MA, Swerdlow NR. Human studies of prepulse inhibition of startle: normal subjects, patient groups, and pharmacological studies. Psychopharmacology (Berl). 2001 Jul;156(2-3):234-58. doi: 10.1007/s002130100810. PMID 11549226
- [Background] Hawk LW Jr, Yartz AR, Pelham WE Jr, Lock TM. The effects of methylphenidate on prepulse inhibition during attended and ignored prestimuli among boys with attention-deficit hyperactivity disorder. Psychopharmacology (Berl). 2003 Jan;165(2):118-27. doi: 10.1007/s00213-002-1235-7. Epub 2002 Nov 1. PMID 12417963
- [Background] Feifel D, Minassian A, Perry W. Prepulse inhibition of startle in adults with ADHD. J Psychiatr Res. 2009 Jan;43(4):484-9. doi: 10.1016/j.jpsychires.2008.06.004. Epub 2008 Jul 31. PMID 18674783
- [Background] Hanlon MC, Karayanidis F, Schall U. Intact sensorimotor gating in adult attention deficit hyperactivity disorder. Int J Neuropsychopharmacol. 2009 Jun;12(5):701-7. doi: 10.1017/S1461145708009711. Epub 2008 Dec 2. PMID 19046483
- [Background] Ashare RL, Hawk LW Jr, Shiels K, Rhodes JD, Pelham WE Jr, Waxmonsky JG. Methylphenidate enhances prepulse inhibition during processing of task-relevant stimuli in attention-deficit/hyperactivity disorder. Psychophysiology. 2010 Sep;47(5):838-45. doi: 10.1111/j.1469-8986.2010.01001.x. Epub 2010 Mar 10. PMID 20233343
- [Background] Takahashi H, Hashimoto R, Iwase M, Ishii R, Kamio Y, Takeda M. Prepulse inhibition of startle response: recent advances in human studies of psychiatric disease. Clin Psychopharmacol Neurosci. 2011 Dec;9(3):102-10. doi: 10.9758/cpn.2011.9.3.102. Epub 2011 Dec 31. PMID 23429840
- [Background] Sable JJ, Kyle MR, Knopf KL, Schully LT, Brooks MM, Parry KH, Diamond RE, Flink LA, Stowe R, Suna E, Thompson IA. The Sensory Gating Inventory as a potential diagnostic tool for attention-deficit hyperactivity disorder. Atten Defic Hyperact Disord. 2012 Sep;4(3):141-4. doi: 10.1007/s12402-012-0079-1. Epub 2012 May 27. PMID 22644992
- [Background] Schulz-Juergensen S, Thiemann A, Gebhardt J, Baumgarten-Walczak A, Eggert P. Prepulse inhibition of acoustic startle and the influence of methylphenidate in children with ADHD. J Atten Disord. 2014 Feb;18(2):117-22. doi: 10.1177/1087054712448960. Epub 2012 Jun 19. PMID 22713361
- [Background] Holstein DH, Vollenweider FX, Geyer MA, Csomor PA, Belser N, Eich D. Sensory and sensorimotor gating in adult attention-deficit/hyperactivity disorder (ADHD). Psychiatry Res. 2013 Jan 30;205(1-2):117-26. doi: 10.1016/j.psychres.2012.08.013. Epub 2012 Sep 25. PMID 23017654
- [Background] Kohl S, Heekeren K, Klosterkotter J, Kuhn J. Prepulse inhibition in psychiatric disorders--apart from schizophrenia. J Psychiatr Res. 2013 Apr;47(4):445-52. doi: 10.1016/j.jpsychires.2012.11.018. Epub 2013 Jan 1. PMID 23287742
- [Background] Feldman HM, Reiff MI. Clinical practice. Attention deficit-hyperactivity disorder in children and adolescents. N Engl J Med. 2014 Feb 27;370(9):838-46. doi: 10.1056/NEJMcp1307215. No abstract available. PMID 24571756
- [Background] Gebhardt J, Schulz-Juergensen S, Eggert P. Maturation of prepulse inhibition (PPI) in childhood. Psychophysiology. 2012 Apr;49(4):484-8. doi: 10.1111/j.1469-8986.2011.01323.x. Epub 2011 Dec 16. PMID 22176532
- [Background] Swerdlow NR, Braff DL, Geyer MA. Cross-species studies of sensorimotor gating of the startle reflex. Ann N Y Acad Sci. 1999 Jun 29;877:202-16. doi: 10.1111/j.1749-6632.1999.tb09269.x. PMID 10415651
- [Background] Grim PF. A sustained attention comparison of children and adults using reaction time set and the GSR. J Exp Child Psychol. 1967 Mar;5(1):26-38. doi: 10.1016/0022-0965(67)90074-4. No abstract available. PMID 6038515
- [Background] Okkesim S, Kara S, Kaya MG, Asyali MH. Analysis of coronary angiography related psychophysiological responses. Biomed Eng Online. 2011 Aug 11;10:71. doi: 10.1186/1475-925X-10-71. PMID 21834993
- [Background] Kumari V, Fannon D, Geyer MA, Premkumar P, Antonova E, Simmons A, Kuipers E. Cortical grey matter volume and sensorimotor gating in schizophrenia. Cortex. 2008 Oct;44(9):1206-14. doi: 10.1016/j.cortex.2007.11.007. Epub 2008 Jan 20. PMID 18761134
- [Background] Molina V, Montes C, Tamayo P, Villa R, Osuna MI, Perez J, Sancho C, Lopez-Albuquerque T, Cardoso A, Castellano O, Lopez DE. Correlation between prepulse inhibition and cortical perfusion during an attentional test in schizophrenia. A pilot study. Prog Neuropsychopharmacol Biol Psychiatry. 2009 Feb 1;33(1):53-61. doi: 10.1016/j.pnpbp.2008.10.011. Epub 2008 Oct 30. PMID 19000732